CLINICAL TRIAL: NCT06962475
Title: A Participant- and Assessor-blinded Superiority Randomized Controlled Trial of Custom Foot Orthoses for Chronic Metatarsalgia
Brief Title: Randomized Controlled Trial of Custom Foot Orthoses for Chronic Forefoot Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2025_UQTR_FOs_RCT
Record Dates: First submitted 2025-01-29; First posted 2025-05-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Metatarsalgia
Keywords: RCT; Metatarsalgia; Foot Orthoses; Sham; Customized
MeSH Terms: conditions — Metatarsalgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants randomized to the intervention group will receive customized FOs for both feet.
  Interventions: Other: Podiatric advice; Other: Customized foot orthoses
- Control group (Sham Comparator): Participants randomized to the control group will receive sham FOs for both feet.
  Interventions: Other: Podiatric advice; Other: Sham foot orthoses

INTERVENTIONS:
Other: Podiatric advice — A podiatrist with 11 years of clinical experience will take the negative foot impressions using a semi-weightbearing method with a foam box for both groups to ensure adequate blinding of participants. Then, the foam boxes of the experimental group will be scanned so that the FOs can be 3D printed. Both groups will receive identical clinical guideline-based information and support at the beginning of the trial. The instructions will be as follows: (1) undertake a familiarization protocol of 14 consecutive full days (2) wear the FOs (customized or sham) at all time when they are standing (targeted minimum of 5 hours per day), (3) avoid positions that cause the metatarsophalangeal joints to dorsiflex (e.g., squatting or tiptoeing), (4) mechanical stress load management according to the tissue stress model, (5) do not walk barefoot and (6) wear shoes with good cushioning in which the FOs will be properly placed.
Other: Customized foot orthoses — The customized foot orthoses will be manufactured with a Nylon-11 shell with 6° medially wedged forefoot-rearfoot posts (2.6 mm if the participants' weight (PW) is inferior or equal to 45 kg; 3.2 mm if 45<PW<100 kg; 4.0 mm if PW>100 kg), a full-length 3 mm Poron top cover and a metatarsal pad (15 shore A) located 5 mm proximal to the metatarsal heads.
  Arms: Intervention Group
Other: Sham foot orthoses — The molded sham FOs will be manufactured from 3 mm ethylene vinyl acetate. They will have an identical top cover material, color and a similar shape than the customized FOs, however, they will provide negligible mechanical support, considering the very low stiffness of their medial arch. The only impact of these FOs on plantar pressure is under the heel. These devices have been used as a sham condition in previous trials and a study has validated them as being credible.
  Arms: Control group

SUMMARY:
Background Chronic metatarsalgia (CM) causes significant pain and disability, affecting quality of life. Foot orthoses (FOs) including medially wedged designs with a metatarsal pad decrease excessive plantar pressure under the metatarsal heads, which is a suggested risk factor for developing CM. This FOs model may be effective in diminishing pain and improving function in these individuals. Thus, the objective of this trial will be to compare the effects of medially wedged FOs with a metatarsal pad and sham FOs on pain and foot function in individuals with CM.

Methods/design This participant- and assessor-blinded superiority randomized controlled trial (RCT) with two parallel groups will be conducted in Trois-Rivières, Canada. Sixty-four participants with CM will be recruited from the Université du Québec à Trois-Rivières outpatient podiatry clinic and via social media invitations. They will be randomized into intervention (customized FOs) or control (sham FOs) groups and will be evaluated at baseline and after 6 and 12 weeks. The primary outcome will be: (1) mean pain during walking for the most painful foot during the past week. The secondary outcomes will be: (1) Foot Function Index, (2) Global rating of change and (3) the 5-level EQ-5D.

Discussion Medially wedged FOs with a metatarsal pad are expected to provide a greater reduction in pain and improvement in foot function compared to sham FOs. This trial will help guide FOs prescription recommendations for managing foot pain in individuals with CM in the future.

DETAILED DESCRIPTION:
Foot musculoskeletal disorders cause significant impairments and disabilities for those affected. Among the various types of foot pain, chronic metatarsalgia (CM) is the most prevalent. Metatarsalgia represents 88% of all causes of foot pain, with a prevalence of 13 to 36% in adults. It is characterized by persistent pain to one or more metatarsophalangeal joints, resulting from harm (whether of mechanical origin or not) to the anatomical structures associated with the joint, including bone, cartilage, capsule and ligaments, tendons, bursae and subcutaneous tissue, and skin. Chronic metatarsalgia significantly reduces the quality of life of those affected, physically, psychologically, and socially. Different treatment modalities are used for CM, such as stretching exercises, footwear modifications, and foot orthoses (FOs). The first-line treatment is conservative, and surgery should be considered only when conservative treatment fails. Nevertheless, there is little high-level evidence (level I) to support the efficacy of conservative treatments for CM.

The reduction of the mechanical overload under the metatarsal heads during locomotion is a fundamental aspect of CM treatment, and it strongly correlates with pain reduction. Foot orthoses are commonly used devices to reduce pain and improve function in individuals with musculoskeletal disorders. They reduce forefoot plantar pressure during locomotion in individuals with CM and redistribute plantar pressure more evenly. Metatarsal pads, a common FOs modification, effectively redistribute forefoot plantar pressure and thus reduce pain caused by excessive metatarsal loads. Adding a medial wedge to FOs (inclination in the frontal plane) further reduces forefoot peak pressure in healthy adults. While FOs tested so far are generally effective in managing CM, their effects can be inconsistent across patients, some patients did not find them effective. From a biomechanical standpoint, FOs reduce mechanical overload; however, it is crucial to determine whether they also effectively reduce pain and improve foot function. Randomized controlled trials (RCT) are considered the gold standard for evaluating treatment effectiveness and efficiently translating research findings into clinical practice. This study design will allow us to assess whether, in addition to their biomechanical effects, FOs provide clinical benefits for individuals with CM.

All details are here : https://doi.org/10.1371/journal.pone.0340905

ELIGIBILITY:
Inclusion Criteria:

1. are aged 18 years or over,
2. have bilateral or unilateral metatarsalgia under one or more of the lesser metatarsal heads for at least 3 months (pain score of ≥ 4 out of 10 on a Visual Analogue Scale (VAS)) that is aggravated by weight-bearing activities,
3. are able to walk without assistive devices (e.g., cane, walker),
4. are willing to wear shoes that will accommodate their FOs on a daily basis and
5. are willing to minimize the use of other interventions (e.g., pain medications, physical therapy) during the trial period

Exclusion Criteria:

1. have arthritis,
2. have neurological diseases (e.g., intermetatarsal neuroma) or other mechanical pain, plantar corns (e.g., intractable plantar keratoma),
3. have a history of orthopedic foot surgery,
4. have prior use of customized FOs,
5. have cognitive impairments,
6. are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Mean pain during walking for the most painful foot during the past week | From Baseline to the end of follow-up at 12 weeks
  visual analog scale (from 0 to 10, 0 being no pain and 10 pain as bad as it could be).

SECONDARY OUTCOMES:
Foot Function Index (FFI) | From Baseline to the end of follow-up at 12 weeks
  The FFI is a widely used, valid, and reliable self-administered questionnaire consisting of 23 items grouped into 3 domains: foot pain (9 items), disability (9 items), and activity limitation (5 items) : we used disability (min: 0, max: 90) and activity limitation (min: 0, max: 50) subscales.
Global rating of change (GROC) | During the follow-up: 6weeks and 12 weeks
  participants' perception of overall treatment effect will be measured using the self-reported global rating of change scale [33]. This outcome will then be dichotomized into the categories of "effective" ("a very great deal better", "a great deal better", "a good deal better" and "moderately better") and "ineffective" ("somewhat better", "a little better", "about the same, hardly any better at all", "no change", "about the same, hardly any worse at all", "a little worse", "somewhat worse", "moderately worse", "a good deal worse", "a great deal worse" and 'a very great deal worse")
Health-related quality of life (HRQoL) | From Baseline to the end of follow-up at 12 weeks
  the 5-level EQ-5D (EQ-5D-5L) will be used [35]. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The participant will be asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

OTHER OUTCOMES:
Demographic and clinical data | Baseline
  Gender: Male, female, non-binary, transgender or other. Age: in years (from the date of birth) Weight: in kg (measured in clinic) Height: in meters (measured in clinic) Body Mass Index: will be calculated with the formula weight divided by height squared Foot Posture Index: The six clinical criteria used in FPI are: 1. Palpation of the talus head (medial and lateral deviation of the talus head in relation to the navicular bone); 2. Curvature of the supra and lateral inframaleolar region; 3. Position of the calcaneus in the frontal plane; 4. Prominence of the talonavicular region; 5. Congruence of the internal longitudinal arche; and 6. Abduction/adduction of the forefoot with respect to the rearfoot. Each criterion is rated between -2 and +2 and the sum of all gives a total score indicating the foot posture (Normal = 0 to +5; pronated = +6 to +9; highly pronated = +10 to +12; supinated = -1 to -4 and highly supinated = -5 to -12).
Effects of the FOs on plantar pressure | Baseline
  peak plantar pressure during a stance phase (kPa) under the metatarsal heads, measured with a Pedar-X in-shoe pressure measurement system (Novel Corporation, Munich, Germany) with foot orthoses and with shod.

CONTACTS AND LOCATIONS:
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Payen Schalkens E, Acien M, Marchand AA, Isabelle PL, Abboud J, Moisan G. Custom foot orthoses for chronic metatarsalgia: Study protocol for a participant- and assessor-blinded superiority randomized controlled trial. PLoS One. 2026 Jan 16;21(1):e0340905. doi: 10.1371/journal.pone.0340905. eCollection 2026. PMID 41544006